CLINICAL TRIAL: NCT01742338
Title: Determining Optimal Dose of Corticosteroids in COPD Exacerbations: A Pilot Study
Brief Title: Dose of Corticosteroids in COPD
Acronym: DOSE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of research staff to recruit participants
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Jeffrey L Carson, MD, Professor of Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0220120019
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Results first posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-03

CONDITIONS: COPD
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Chronic bronchitis; emphysema; Corticosteroids
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Emphysema | interventions — Adrenal Cortex Hormones; Prednisone; Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low Dose Corticosteroids (Active Comparator): 10 mg IV q8hrs x 3 days*, then prednisone 40 mg PO daily x 4 days, then prednisone 30 mg daily x 1 day, then prednisone 20 mg daily x 1 day, then prednisone 10 mg daily x 1 day, then stop.
  *If patient unable to receive IV medications, will give prednisone 20 mg PO bid for the first 3 days.
  Interventions: Drug: Low Dose Corticosteroids
- High Dose Corticosteroids (Experimental): Methylprednisolone 40 mg IV q8hrs x 3 days*, then prednisone 80 mg PO daily x 4 days, then prednisone 60 mg daily x 1 day, then prednisone 40 mg daily x 1 day, then prednisone 20 mg daily x 1 day, then stop. *If patient unable to receive IV medications, will give prednisone 40 mg PO bid for the first 3 days.
  Interventions: Drug: High Dose Corticosteroids

INTERVENTIONS:
Drug: Low Dose Corticosteroids
  Other Names: prednisone; methylprednisolone; Solumedrol
  Arms: Low Dose Corticosteroids
Drug: High Dose Corticosteroids
  Other Names: prednisone; methylprednisolone; Solumedrol
  Arms: High Dose Corticosteroids

SUMMARY:
COPD (chronic obstructive pulmonary disease) is a long-lasting lung disease usually caused by long-term smoking. COPD can get worse, making people sick enough to need hospitalization. Corticosteroids are very effective and are almost always used, but nobody knows the right dose. High doses may work better but could cause more side effects than low doses. Typical treatment lengths last at least one week. This study will be comparing two common regimens: either 40mg of corticosteroids daily (low dose), or 80mg of corticosteroids daily (high dose). It is unknown which regimen works better..

DETAILED DESCRIPTION:
The goal of the study is to determine whether a high-dose corticosteroid regimen in patients admitted to the hospital with COPD exacerbations is associated with better clinical outcomes and at acceptable risk of adverse effects compared to a low-dose corticosteroid regimen. Our hypothesis is that high-dose corticosteroids is associated with a decreased rate of treatment failure, shorter length of hospital stay, and improved quality of life with similar risk of adverse effects. The study population includes patients ≥ 40 years-old with a ≥ 10 pack-years smoking history and a diagnosis of COPD, emphysema, or chronic bronchitis who present to the emergency room with increased dyspnea, increased sputum, or increased cough that requires admission to the hospital. We will perform a prospective, randomized, double-blinded study to determine if a high-dose corticosteroid regimen, which is already in use in clinical practice, decreases treatment failure compared to a low-dose corticosteroid regimen that is based on national consensus guidelines.

ELIGIBILITY:
Inclusion Criteria:

i. Patients with a diagnosis of COPD, emphysema, or chronic bronchitis ii. Age ≥ 40 years-old iii. Smoking history ≥ 10 pack-years iv. Presentation to the emergency room with increased dyspnea, increased sputum, or increased cough v. Admission to the hospital

Exclusion Criteria:

i. Alternative diagnosis for cause of dyspnea, increased sputum or cough ii. Patients who requires intubation at time of recruitment iii. Patients who are unable to give consent iv. Patients who are pregnant or could be pregnant or are currently breast-feeding v. Women of child-bearing age who cannot use methods of contraception as described in the consent, including condoms, female condoms, cervical caps, diaphragms, and intra uterine devices.

vi. Patients who were previously entered into the trial and are re-admitted to the hospital with a new COPD exacerbation.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Carson, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (2):
- United States (2):
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University Medical Center at Princeton, Plainsboro, New Jersey

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Corticosteroids: 10 mg IV q8hrs x 3 days*, then prednisone 40 mg PO daily x 4 days, then prednisone 30 mg daily x 1 day, then prednisone 20 mg daily x 1 day, then prednisone 10 mg daily x 1 day, then stop.
  *If patient unable to receive IV medications, will give prednisone 20 mg PO bid for the first 3 days.
  Low Dose Corticosteroids
- High Dose Corticosteroids: Methylprednisolone 40 mg IV q8hrs x 3 days*, then prednisone 80 mg PO daily x 4 days, then prednisone 60 mg daily x 1 day, then prednisone 40 mg daily x 1 day, then prednisone 20 mg daily x 1 day, then stop. *If patient unable to receive IV medications, will give prednisone 40 mg PO bid for the first 3 days.
  High Dose Corticosteroids
Period: Overall Study
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids
Started | 47 | 42
Completed | 43 | 39
Not Completed | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids | Total
Number analyzed (Participants) | 47 | 42 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (11.3) | 65.9 (10.3) | 65.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 19 | 40
  Male | 26 | 23 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 7 | 20
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment Failure
Description: Composite outcome of treatment failure defined as death, intubation, re-admission for COPD exacerbation, or intensification of therapy (increased steroid use, change of antibiotic therapy) within a 30-day follow-up period.
Time Frame: 30 days
Population: Data available for 43 participants the Low Dose Arm and 39 participants in the High Dose Arm
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids
Number analyzed (Participants) | 43 | 39
Participants | 14 | 10

2. Secondary Outcome: Length of Stay
Description: Hospital days from randomization to discharge
Time Frame: 30 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids
Number analyzed (Participants) | 47 | 42
days | 2 [0 to 3] | 2 [1 to 4]

3. Secondary Outcome: Quality of Life Score
Description: Quality of life measured by Clinical COPD Questionnaire. The Clinical COPD Questionnaire consists of 10 questions about the severity of COPD symptoms and limitation of activities over the prior week.
Time Frame: 30 days
Population: Data are missing for 6 in the Low Dose Arm and 5 in the High Dose Arm
Measure: Median (Inter-Quartile Range); unit: score on scale of 0 (best) to 6 (worst)
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids
Number analyzed (Participants) | 41 | 37
score on scale of 0 (best) to 6 (worst) | 1.8 [0.8 to 2.8] | 1.8 [1.2 to 2.7]

4. Other Pre Specified Outcome: Adverse Effects
Description: Composite outcome of short-term adverse effects. Defined as hyperglycemia, hypertension, adrenal suppression, psychiatric disturbance, infection, and gastrointestinal bleed that require a consultation, an invasive procedure, or initiation of a specific therapy.
Time Frame: 30 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 Days
Description: Data are missing for 1) Death - 5 in the Low Dose Arm; 2 in the High Dose Arm 2) COPD Exacerbation - 5 in the Low Dose Arm; 3 in the High Dose Arm 3) Theraputic Intensification - 4 in the Low Dose Arm; 3 in the High Dose Arm
Arm/Group | Low Dose Corticosteroids | High Dose Corticosteroids
All-Cause Mortality (participants affected / at risk) | 0/42 | 1/40
Serious Adverse Events (participants affected / at risk) | 2/42 | 2/39
Other Adverse Events (participants affected / at risk) | 12/43 | 10/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Corticosteroids (N=42) | High Dose Corticosteroids (N=39)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) — COPD exacerbation requiring admission to the hosptial
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Corticosteroids (N=43) | High Dose Corticosteroids (N=39)
Theraputic Instensification (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 10 (10) — Required additional or increased dosage of medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT01742338/Prot_SAP_000.pdf
  • Informed Consent Form (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT01742338/ICF_001.pdf